CLINICAL TRIAL: NCT05726812
Title: A Group Training to Plan and Organize for Adolescents With ADHD: Effectiveness and Feasibility
Brief Title: Plan My Life Together; a Group Training for Adolescents With ADHD
Status: Completed | Type: Observational
Sponsor: GGZ Noord-Holland-Noord (Other)
Collaborators: Universiteit Leiden (Other)
Responsible Party: Sponsor
Other Study IDs: GGZNHN
Record Dates: First submitted 2022-12-09; First posted 2023-02-14 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: ADHD; Adolescence
Keywords: Planning and organization skills; Plan My Life; Group Training
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Plan My Life Together — A group training for adolescents with ADHD in which they learn to plan and organize. The training consists of 8 weekly sessions of 90 minutes for the adolescent and 2 parent sessions of 90 minutes.

SUMMARY:
This observational study is a first orientation on the effects and feasibility of a group training to plan and organize for adolescents with attention deficit disorder (ADHD). This study focuses on the following questions:

* Is there an improvement on planning skills after training?
* Are there fewer ADHD characteristics after training?
* Is there an improvement on self-esteem after training?
* How feasible is a group training for adolescents with ADHD?
* How satisfied are practitioners and adolescents about the training?

Based on the effect-size of the individual training variant, the literature on the effect of group treatment and the adolescent target group, in which the peer group gets more important, the hypothesis is that the group training Plan My Life Together will have a medium to large effect on planning skills. Furthermore, positive effects on ADHD characteristics and self-esteem are also expected. The assumption is that Plan My Life Together is feasible and suitable.

DETAILED DESCRIPTION:
Attention deficit and/or hyperactivity and impulsivity disorder (ADHD) has a high prevalence in the adolescence. In this age stage, where independence and personal responsibility become increasingly important, ADHD is characterized mainly by problems in executive functions and there are often problems in planning schoolwork.This is frequently accompanied by tensions in the family. More co-morbidity also develops, including problems in self-image, as a result of negative feedback from the environment. Individual behavioral treatment has been found to be effective in reducing ADHD symptoms. In the ADHD guidelines (cognitive) behavioral therapy aimed at planning and organization, with consideration for motivational interviewing elements, is recommended for adolescents.

In the individual training Plan My Life, adolescents learn to plan their school and homework better through cognitive behavioral therapy (CBT) and motivational interviewing, so that they have fewer problems with their ADHD characteristics and have more positive experiences. The training is proven effective, few adolescents drop out, and parents and practitioners are positive about the training. The training was developed and studied on an individual basis.

There may be advantages to offering this training in a group setting. Among other things, the group can serve as a catalyst and experiences can be shared. Group therapy has been shown to work for several mental disorders, in some cases even better than the individual therapy. It is obvious that in adolescence the group is relatively even more important. Also, group treatment can be more efficient.

ELIGIBILITY:
Inclusion Criteria:

* adolescents with an ADHD classification according to the DSM-5.
* age 12 to 16 years.
* outpatient treatment at "GGZ-NHN" (specialized mental health care service in the Netherlands)) or at "Psychologenpraktijk Kuin" (first-line psychological mental health care, Haarlem)
* currently following secondary regular education
* Intention to participate in the group and willingness to fill out questionnaires several times.

Exclusion Criteria:

* a DSM-5 classification of autism
* acute crisis situation (acute suicidality, acute psychotic symptoms, addiction problems requiring immediate treatment, or unsafe home situation)
* Insufficient mastery of the Dutch language.

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Participants are from the region "North-Holland" and receive mental health care for ADHD and possible other mental health problems. Medication use is allowed if participants function stable on medication.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-07-15 (Actual)

PRIMARY OUTCOMES:
Change in the subscale scores plan/organize - self rated (from BRIEF-2, see description)) | Baseline (start study) - T0 (=9 weeks after start study, intervention starts) - T1 (=18 weeks after start study) - T2 (=27 weeks after start study)
  Subscale plan/organize from the Behavior Rating Inventory of Executive Function - Adolescent version
  Higher scores indicated better planning/organizing scales. Subscale ranges from 8 - 24
Change in the subscale score plan/organize - parent rated (from BRIEF-2, see description) | Baseline (start study) - T0 (=9 weeks after start study, intervention starts) - T1 (=18 weeks after start study) - T2 (=27 weeks after start study)
  Subscale plan/organize from the Behavior Rating Inventory of Executive Function - Parent version
  Higher scores indicated better planning/organizing scales. Subscale ranges from 8 - 24

SECONDARY OUTCOMES:
Change in AVL - parent rated (see description) | Baseline (start study) - T0 (=9 weeks after start study, intervention starts) - T1 (=18 weeks after start study) - T2 (=27 weeks after start study)
  ADHD Vragenlijst - ouders (ADHD rating scale, Dutch version)
  Higher scores indicate more ADHD-symptoms. Range: 0 - 72
Change in RSES - self rated (see description) | Baseline (start study) - T0 (=9 weeks after start study, intervention starts) - T1 (=18 weeks after start study) - T2 (=27 weeks after start study)
  Rosenberg Self Esteem Scale - Adolescent version
  Higher scores indicate more self-esteem. Range: 0-40
Change in RSES - parent rated (see description) | Baseline (start study) - T0 (=9 weeks after start study, intervention starts) - T1 (=18 weeks after start study) - T2 (=27 weeks after start study)
  Rosenberg Self Esteem Scale - Parent version
  Higher scores indicate more self-esteem. Range: 0-40

OTHER OUTCOMES:
Scale questions on satisfaction | Only at T2 (=27 weeks after start study)
  Scale questions for practitioners and adolescents to measure satisfaction with the group training
  Higher scores indicate more satisfaction. Range: 1-10.

CONTACTS AND LOCATIONS:
Overall Officials: Manon van Hensbergen, MSc, Principal Investigator — GGZ Noord-Holland-Noord
Locations (1):
- GGZ Noord-Holland-Noord, Heerhugowaard, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
Anonimized data will be shared upon request and careful consideration of research plan by the principal investigators.